CLINICAL TRIAL: NCT07274332
Title: Acute Effects of Different Frequencies of Auricular Vagus Nerve Stimulation on HRV, Blood Pressure, and Respiratory Rate: A Sham-Controlled, Randomized, Crossover Dose-Response Study
Brief Title: Frequency-Dependent Effects of Auricular Vagus Nerve Stimulation on Autonomic and Cardiovascular Parameters
Acronym: AVNS-DRC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SEFA HAKTAN HATIK (Other)
Responsible Party: Sponsor-Investigator, SEFA HAKTAN HATIK, Assistant Professor, Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: tcVNS1; IRB Number (Pending) (Registry Identifier: Gümüşhane University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Vagus Nerve Stimulation; Autonomic Nervous System; Heart Rate; Blood Pressure; Respiration; Healthy Volunteers
Keywords: Transcutaneous Cervical Vagus Nerve Stimulation; Neuromodulation; Non-invasive Vagus Stimulation; Parasympathetic Activation; Heart Rate Variability
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: All participants receive each of the five stimulation conditions in randomized counterbalanced order (Williams Latin Square). Each visit includes a 10-minute tcVNS session and before/after physiological recordings. Washout between visits is ≥48 hours.
Who Masked: Participant
Masking Description: Participants are blinded to the stimulation condition. The Pulsetto FIT™ device displays active lights and interface indicators in both sham and active frequencies, but delivers no current in the sham arm (0 Hz).
  The investigator administering the stimulation is aware of the condition due to device programming requirements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1 - Sham (0 Hz) (Sham Comparator): Intervention Type: Pulsetto FIT™ tcVNS Device Intervention Name: Sham tcVNS Description: Device placed on bilateral cervical region; no electrical current delivered.
  Dose: 10 minutes
  Interventions: Device: Pulsetto FIT™ - Sham tcVNS
- 2 - 10 Hz tcVNS (Experimental): Intervention Type:Pulsetto FIT™ tcVNS Device Intervention Name: tcVNS (10 Hz) Description: Bilateral cervical stimulation at 10 Hz, 250 μs pulse width. Duration: 10 minutes
  Interventions: Device: Pulsetto FIT™ - tcVNS 10 Hz
- 3 - tcVNS 25 Hz (Experimental): Intervention Type:Pulsetto FIT™ tcVNS Device Intervention Name: tcVNS (25 Hz) Description: Bilateral cervical stimulation at 25 Hz, 250 μs pulse width. Duration: 10 minutes
  Interventions: Device: Pulsetto FIT™ - tcVNS 25 Hz
- 4 - tcVNS 50 Hz (Experimental): Intervention Type:Pulsetto FIT™ tcVNS Device Intervention Name: tcVNS (50 Hz) Description: Bilateral cervical stimulation at 50 Hz, 250 μs pulse width. Duration: 10 minutes
  Interventions: Device: Pulsetto FIT™ - tcVNS 50 Hz
- 5 - tcVNS 100 Hz (Experimental): Intervention Type:Pulsetto FIT™ tcVNS Device Intervention Name: tcVNS (100 Hz) Description: Bilateral cervical stimulation at 100 Hz, 250 μs pulse width. Duration: 10 minutes
  Interventions: Device: Pulsetto FIT™ - tcVNS 100 Hz

INTERVENTIONS:
Device: Pulsetto FIT™ - Sham tcVNS — The Pulsetto FIT™ device is placed bilaterally on the cervical region (posterior margin of the sternocleidomastoid muscle).
  In the sham condition, the device displays normal operational lights but delivers no electrical stimulation (0 Hz; inactive mode).
  This condition is used for blinding and as the control comparator. Dose: 10 minutes
  Arms: 1 - Sham (0 Hz)
Device: Pulsetto FIT™ - tcVNS 10 Hz — Bilateral transcutaneous cervical vagus nerve stimulation delivered via the Pulsetto FIT™ device at 10 Hz, 250 µs pulse width.
  Current intensity adjusted to a mild, non-painful tingling sensation, individualized for each participant.
  Dose: 10 minutes
  Arms: 2 - 10 Hz tcVNS
Device: Pulsetto FIT™ - tcVNS 25 Hz — Bilateral tcVNS using the Pulsetto FIT™ device at 25 Hz, 250 µs pulse width. Stimulation intensity set at a comfortable sensory level. Dose: 10 minutes
  Arms: 3 - tcVNS 25 Hz
Device: Pulsetto FIT™ - tcVNS 50 Hz — Bilateral cervical vagus nerve stimulation via Pulsetto FIT™ at 50 Hz, 250 µs pulse width.
  Intensity adjusted to a tolerable sensory level without discomfort. Dose: 10 minutes
  Arms: 4 - tcVNS 50 Hz
Device: Pulsetto FIT™ - tcVNS 100 Hz — Bilateral tcVNS delivered with the Pulsetto FIT™ device at 100 Hz, 250 µs pulse width.
  Highest stimulation frequency used in this protocol; current intensity individualized per participant comfort.
  Dose: 10 minutes
  Arms: 5 - tcVNS 100 Hz

SUMMARY:
This randomized, sham-controlled, crossover study investigates the acute autonomic effects of transcutaneous cervical vagus nerve stimulation (tcVNS) applied at five different frequencies (0 Hz/sham, 10 Hz, 25 Hz, 50 Hz, 100 Hz) in healthy adults. The primary objective is to determine how stimulation frequency modulates heart rate variability (HRV), blood pressure, and respiratory rate. The study aims to establish a frequency-specific dose-response model using validated physiological measurements.

DETAILED DESCRIPTION:
Transcutaneous cervical vagus nerve stimulation (tcVNS) is a non-invasive neuromodulation technique capable of activating afferent vagal pathways projecting to autonomic brainstem nuclei. Although previous studies demonstrate tcVNS-related modulation of autonomic functions, the frequency-response relationship remains insufficiently explored.

This crossover trial randomizes participants to receive five stimulation conditions (sham, 10 Hz, 25 Hz, 50 Hz, 100 Hz) in counterbalanced order. HRV (Polar H10), blood pressure (Omron), and respiratory rate (Kinovea-based thoracoabdominal video tracking) are collected pre- and post-stimulation. Washout between sessions is ≥48 hours.

The study provides one of the first systematic evaluations of frequency-dependent tcVNS effects in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years
* Healthy (self-reported)
* No cardiovascular, neurological, metabolic or psychiatric disorders
* No regular medication affecting autonomic function
* Non-smoker
* BMI 18-29.9

Exclusion Criteria:

* Pregnancy
* Cardiac arrhythmia
* Hypertension or hypotension
* Chronic respiratory disorders
* Active infection
* Metal implants in cervical area
* Epilepsy
* Syncope history
* Prior vagus stimulation experience

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) Changes (ΔRMSSD, ΔHF, ΔLF/HF) | Pre- vs Post-stimulation (5-min segments)(5-minute baseline, 5-minute stimulation, 5-minute post period)
  HRV is recorded using a validated high-resolution heart rate monitor (Polar H10) during a 5-minute resting baseline (T0) and a 5-minute post-stimulation period (T2).
  The following time- and frequency-domain parameters are analyzed: RMSSD, HF (ms²), and LF/HF ratio.
  Artefact correction is performed using standard HRV processing methods. Acute autonomic response is quantified by calculating change scores (Δ = post-pre) for each stimulation frequency.

SECONDARY OUTCOMES:
Blood Pressure (SBP, DBP, MAP) | Pre- vs Post-stimulation (5-minute baseline, 5-minute stimulation, 5-minute post period)
  Two readings are taken at each time point from the right arm with a validated automatic sphygmomanometer, and the average systolic, diastolic, and mean arterial pressure values are used for analysis.
  Changes are calculated as post-pre (Δ values) to assess the acute physiological effect of each stimulation frequency..
Respiratory Rate (breaths per minute) | Pre- vs Post-stimulation (5-minute video segments) (5-minute baseline, 5-minute stimulation, 5-minute post period)
  Respiratory rate is assessed by video-based thoracoabdominal motion tracking at baseline (T0) and after stimulation (T2).
  Videos are analyzed using Kinovea motion-tracking software, and a 1-minute stable segment is used to determine breaths per minute by counting inspiratory peaks.
  Respiratory changes are expressed as Δ values (post-pre) to account for individual differences and improve HRV interpretability.Respiratory rate is assessed by video-based thoracoabdominal motion tracking at baseline (T0) and after stimulation (T2).
  Videos are analyzed using Kinovea motion-tracking software, and a 1-minute stable segment is used to determine breaths per minute by counting inspiratory peaks.
  Respiratory changes are expressed as Δ values (post-pre) to account for individual differences and improve HRV interpretability.
Discomfort Level (Visual Analog Scale, 0-10) | Pre- vs Post-stimulation (5-minute baseline, 5-minute stimulation, 5-minute post period)
  Participants report their perceived discomfort level at baseline (T0) and immediately after stimulation (T2) using a 0-10 Visual Analog Scale (VAS).
  The scale captures any sensory discomfort associated with tcVNS. Changes are calculated by subtracting the pre-stimulation score from the post-stimulation score (ΔVAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Sinop University, Türkeli Vocational School (Türkeli MYO), Türkeli, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study includes physiological recordings (HRV, blood pressure, respiratory videos) that cannot be fully anonymized. Data sharing may pose a risk of indirect identification.
  Only aggregated results will be reported in publications and presentations.
  IPD Sharing Time Frame:
  Not applicable.
  IPD Sharing Access Criteria:
  Not applicable.

REFERENCES:
- [Result] Kranz S, Lukacs J, Bishop J, Block ME. Intergeneration transfer of diet patterns? Parental self-report of diet and their report of their young adult children with ASD. PLoS One. 2022 Feb 8;17(2):e0263445. doi: 10.1371/journal.pone.0263445. eCollection 2022. PMID 35134082
- [Result] Alsoufi B. Curb Your Enthusiasm for the Ozaki Procedure in Small Children. Ann Thorac Surg. 2022 Jan;113(1):378-379. doi: 10.1016/j.athoracsur.2021.03.085. Epub 2021 Apr 8. No abstract available. PMID 33839137
- [Result] Nordahl HM, Wells A. Metacognitive Therapy of Early Traumatized Patients With Borderline Personality Disorder: A Phase-II Baseline Controlled Trial. Front Psychol. 2019 Jul 30;10:1694. doi: 10.3389/fpsyg.2019.01694. eCollection 2019. PMID 31417453
- [Result] Peuker ET, Filler TJ. The nerve supply of the human auricle. Clin Anat. 2002 Jan;15(1):35-7. doi: 10.1002/ca.1089. PMID 11835542
- [Result] Grossman P, Taylor EW. Toward understanding respiratory sinus arrhythmia: relations to cardiac vagal tone, evolution and biobehavioral functions. Biol Psychol. 2007 Feb;74(2):263-85. doi: 10.1016/j.biopsycho.2005.11.014. Epub 2006 Nov 1. PMID 17081672
- [Result] Zhang Y, Xiao S, Feng H, Zhang L, Zhou Z, Hu W. Self-interference cancellation using dual-drive Mach-Zehnder modulator for in-band full-duplex radio-over-fiber system. Opt Express. 2015 Dec 28;23(26):33205-13. doi: 10.1364/OE.23.033205. PMID 26831988
- [Result] Fernandes TL, Viezzer Fernandes B, Jitumori C, Franco GCN. A Case Report of Oral Bisphosphonate Treatment for Osteoporosis Leading to Atypical Femoral Fracture and Pathologic Mandibular Fracture. Am J Case Rep. 2023 Oct 23;24:e941144. doi: 10.12659/AJCR.941144. PMID 37867315